CLINICAL TRIAL: NCT04248647
Title: Surgical Prehabilitation of Cancer Patients Undergoing Colorectal Resection. Modalities to Mitigate the Level of Anxiety and Depression Prior to Surgery.
Brief Title: Surgical Prehabilitation of Cancer Patients Undergoing Colorectal Resection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Franco Carli, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMPI/2017-2840
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Cancer
Keywords: Psychological prehabilitation; Colorectal cancer; Functional capacity; Physical activity; Nutrition; Psychological counselling
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): 4-week multimodal preoperative intervention (i.e., Prehabilitation) consisting of an aerobic and strength training program, nutritional counselling and psychological support to help improve physical and psychological health prior to surgical resection of colorectal cancer.
  Interventions: Behavioral: Multimodal prehabilitation

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — This arm will receive a 4-week prehabilitation program consisting of:
  Exercise: Participants will receive a 3x/week aerobic and strength training exercise program. They will perform 2 workouts per week at home and attend an in-hospital supervised exercise session once per week.
  Nutritional counselling: Participants will meet with a registered dietician who will provide personalized nutritional recommendations and a whey protein supplement, tailored according to participants' self-reported dietary intake and anthropometric measurements.
  Psychological support: Participants will receive a 90-minute session at baseline, and weekly in-hospital follow-ups throughout the preoperative period. The sessions will aim to reduce preoperative distress and improve adherence to the exercise program and nutritional recommendations. Psychological support will be delivered by a trained master's student, under the direct supervision of a registered Clinical Psychologist.

SUMMARY:
Psychological distress is common among adults newly diagnosed with cancer and those awaiting cancer treatment(s). Although preoperative psychological distress has been shown to be associated with poorer physical health and adverse treatments among colorectal cancer survivors, few psychological interventions have been developed to reduce distress, and improve physical health in the preoperative period. Moreover, whether a preoperative psychological intervention, delivered in addition to a multimodal Prehabilitation program can improve psychological and physical health remains unknown. Therefore, the purpose of this pilot cohort study was to examine the impact of a structured psychological intervention, given in addition to standard Prehabilitation, on preoperative psychological health and functional capacity in colorectal cancer patients awaiting surgery.

DETAILED DESCRIPTION:
All participants will receive a multimodal prehabilitation program preoperatively for 4 weeks, composed of three elements: aerobic and strength training exercise program, nutritional counselling and psychological support. The exercise program will be three times per week and include a combination of home-based (twice per week) and supervised (once per week) sessions. Participants' nutritional status and dietary intake will be assessed by a registered dietician/nutritionist, and a whey protein supplement (Immunocal) will be prescribed to achieve a daily intake of 1.5 g protein/kg. Psychological support will consist of a 90-minute interview/session at baseline and weekly in-person follow-ups before surgery aimed at reducing psychological distress and improving adherence to the exercise program and nutritional recommendations. Perioperative care will follow the McGill Surgical Recovery Pathway, also called Enhanced Recovery Program, which is an evidence-based care plan set up by the Surgical Recovery (SuRe) multidisciplinary committee of the McGill University Health Centre.

ELIGIBILITY:
Inclusion Criteria:

* Currently aged 18 years or older
* Diagnosed with non-metastatic, colorectal cancer
* Awaiting resection of malignant colorectal lesions
* Able to provide informed consent in English or in French

Exclusion Criteria:

- Have health condition(s) interfering with ability to safely perform exercise at home or to complete testing procedures (e.g., non-ambulatory, dementia, severe end-organ disease, morbid obesity, cardiac abnormalities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Functional capacity: Six-minute walk test (Enright, 2003) | Baseline (week 0), post-intervention (week 4)
  Change in participants' performance on the six-minute walk test (6MWT) across baseline (week 0), and post-intervention (week 4). The 6MWT measures the distance an individual can walk, in metres, in a 6-minute period. Greater distance walked during the 6MWT indicates greater functional capacity.

SECONDARY OUTCOMES:
Postoperative complications: Clavien Classification (Dindo, Demartines & Clavien, 2004) | 8-weeks post-surgery (week 12)
  Postoperative complications (e.g., pneumonia, urinary tract infection, hemorrhage, bile leak) following colorectal resection will be measured and scored using the Clavien Classification. Each complication is graded between I ('Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy') to V ('Death of a patient') with higher grades indicating greater severity of complication.
Depressive and anxiety symptoms: The Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) | Baseline (week 0), post-intervention (week 4)
  Change in participants' self-reported anxiety and depressive symptoms across baseline (week 0), and post-intervention (week 4). Each item is scored on a 0 (e.g., 'Definitely as much') to 4 (e.g., 'Hardly at all') scale with higher scores representing greater severity of anxiety and depressive symptoms.
Health related quality of life: RAND 36-item Short Form Health Survey (SF-36; Ware & Sherbourne, 1992) | Baseline (week 0), post-intervention (week 4)
  Change in participants' self-reported quality of life across baseline (week 0), and post-intervention (week 4). The SF-36 measures eight dimensions: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0-100 scale, with higher scores representing a more favourable health state.
Physical activity: Community Health Activities Model Program for Seniors (CHAMPS; Stewart et al., 2001) | Baseline (week 0), post-intervention (week 4)
  Change in participants' self-reported physical activity levels across baseline (week 0), and post-intervention (week 4). CHAMPS measures the average number of hours individuals report engaging in 41 different activities (or varying intensities) during a typical week. Metabolic equivalent of task (MET) scores are calculated for activities engaged in at mild, moderate and vigorous intensity with higher scores indicating higher levels of engagement.
Lower body strength: Sit-to-Stand test (Bohannon, 1995) | Baseline (week 0), post-intervention (week 4)
  Change in participants' objective performance on the sit-to-stand test across baseline (week 0), and post-intervention (week 4). The sit-to-stand test measures lower body strength by recording the maximum number of times an individual can go from a seated position to a standing position, without using their arms, in a 30-second period.
Nutritional status: body weight loss, serum albumin, hand grip strength, body mass index, lean body mass and percentage of body fat | Baseline (week 0), post-intervention (week 4)
  Change in nutritional status across baseline (week 0), and post-intervention (week 4). Body mass index (kg/m2), lean body mass and percentage of body fat will be measured using a bioimpedance machine. Self-reported body weight loss in the preceding three months will be recorded. Serum albumin will be measured via blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41. doi: 10.1097/00005768-200107000-00010. PMID 11445760
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188